CLINICAL TRIAL: NCT01368367
Title: Safety and Efficacy of Exercise Training Post Burn Injury: a Randomized Controlled Trial
Brief Title: Exercise Training Post Burn Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Queensland (Other)
Collaborators: Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Dr Jennifer Paratz, University of Queensland
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETPB1
Record Dates: First submitted 2011-05-27; First posted 2011-06-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2010-11

CONDITIONS: Burns
Keywords: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive exercise group (Active Comparator)
  Interventions: Other: Intensive exercise
- Stretch exercise only (Placebo Comparator)
  Interventions: Other: Intensive exercise

INTERVENTIONS:
Other: Intensive exercise — Both groups, stretching exercise monitored once per week Intensive exercise group An aerobic and resisted exercise program for a minimum of three times per week for a total of approximately 60 minutes per session for six weeks. Aerobic exercise will be conducted on a treadmill, exercise bike or arm ergometer at an intensity of 80 % of VO2peak during initial assessment. For resistance exercise, the three repetition maximum (3RM) (maximum weight able to be lifted a maximum of 3 times) will be established and then resisted exercise will be commenced at 60% of the 3RM in the first week. Resisted exercise will then be progressed weekly by 5-10% by increasing the number of repetitions or the weights lifted. All resisted exercises will be done using variable resistance machines or free weights.

SUMMARY:
The purpose of this study is to determine whether a high intensity aerobic and resisted exercise program will improve physical, functional and psychological outcomes in patients post burn injury.

DETAILED DESCRIPTION:
Even though immediate and early death from severe thermal injury has reduced over the last twenty years, considerable physical and psychosocial morbidity still persists. While exercise is strongly recommended to assist recovery and overall outcome, there is limited evidence in adults to indicate whether it is effective and/or safe.

This study will investigate the effect of a high intensity aerobic and resisted exercise program exercise program on safety, physical, functional and quality of life measures in adults post burn injury.

ELIGIBILITY:
Inclusion Criteria:

* Burns greater than 20% total body surface area
* 18 years of age and over
* English speaking
* Post final grafting procedure

Exclusion Criteria:

* Accompanying anoxic brain injury
* Cardiac disease or injury (American College of Sports medicine ACSM criteria)
* Quadriplegia
* Severe behaviour or cognitive disorders
* Compassionate care only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2007-12; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Burns Specific Health Scale - Abbreviated (BSHS-A) | Change from baseline to six weeks, change from 6 weeks to 12 weeks
  The BSHS-A is an injury specific self reported questionnaire consisting of 80 questions encompassing four primary domains namely physical, psychological, social and general, with reports of good internal consistency, test/ retest reliability and strong convergent validity data.

SECONDARY OUTCOMES:
The modified shuttle walk test (MSWT) | Change from baseline to six weeks, change from 6 weeks to 12 weeks
  The modified shuttle walk test (MSWT) is an established test of functional exercise capacity. It is an objective measure with 15 incremental levels of both walking and running. Total distance acheived will be recorded.
VO2peak (ie the volume of oxygen consumed by the cells at the most intensive level during the exercise test) | Change from baseline to six weeks, change from 6 weeks to 12 weeks
  VO2peak (ie the volume of oxygen consumed by the cells at the most intensive level during the modified shuttle walk test) will be recorded by a portable metabolic monitor (Metalyzer 3B analyser (Cortex:biophysik, GMbH, Germany) Cortex MetaMax 3B).
Resting heart rate (beats/minute) | Change from baseline to six weeks, change from 6 weeks to 12 weeks
  Resting heart rate was recorded by a polar heart rate monitor (PE3000, Polar Electro, Kemple, Finland) in beats/minute.
Muscle strength | Change from baseline to six weeks, change from 6 weeks to 12 weeks
  Muscle Strength - a baseline measure of the quadriceps and latisimuss dorsi muscles will be taken by the one repetition maximum or 1RM. This is the maximum amount of weight one can lift in a single repetition for a given exercise and has been utilized as an outcome measure in subjects post burns.
Grip strength | Change from baseline to six weeks, change from 6 weeks to 12 weeks
  Grip strength will be measured using a Jamar dynamometer as per the protocol for the American Hand Therapists Society with an average of three measurements taken. This dynamometer is a hydraulic appliance which can measure grip strength in five alternate grip position settings. This has been shown to have good reliability and validity and is considered the gold standard of hand grip measurement.
QuickDash | Change from baseline to six weeks, change from 6 weeks to 12 weeks
  The Quick disabilities of the arm, shoulder and hand (QuickDASH)is a self rated questionnaire on upper limb function with good repeatability, validity and responsiveness in burns patients. Sixty percent of the questions relate to overall upper limb disability with the remainder of the optional questions relating to work, sports and musical activities. Lower scores on this scale indicate less disability of the upper limb.
The Lower Extremity Functional Scale (LEFS) | Change from baseline to six weeks, change from 6 weeks to 12 weeks
  The Lower Extremity Functional Scale (LEFS) measures disability related to the lower extremities with regard to work, activities of daily living and recreation and has been shown to have sensitivity to change in burns patients and excellent test-retest reliability and construct validity in general patients. Higher scores indicate less disability with a possible total of 80.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brisbane & Womens Hospital, Brisbane, Queensland, Australia